CLINICAL TRIAL: NCT00143013
Title: Gene Expression Profiling by DNA Chips and Subsequent Bioinformatic Analysis for Identification of Genes and Biochemical Pathways Associated With Type 2 Diabetes
Brief Title: Gene Expression Profiling and Bioinformatic Analysis Identifying Genes and Biochemical Pathways in Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Other Study IDs: 002
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; microarray; skeletal muscle; bioinformatics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Type 2 diabetes is a disorder of the metabolic system that greatly affects individual health and imposes significant cost for society on health care. It is necessary to initiate research with emphasis on improvement on quality of life and reduce the serious complications as a result of type 2 diabetes.

In type 2 diabetes insulin resistance and impairment of insulin secretion by beta-cells are the major pathophysiological defects and characterized by raised plasma glucose levels. Today, little is known about gene regulation and biochemical pathways involved in the disease.

Bioinformatics and gene expression microarrays (GEM) will be applied to gain insight into the molecular pathophysiology of type 2 diabetes. The simultaneous monitoring of thousands of genes in parallel can identify novel genes and entire biochemical pathways that are dysregulated at the transcriptional level. Affymetrix Inc. chips or spotted arrays will be applied as DNA microarray tools. Bioinformatic software programs and databases will be employed as data mining tools in order to perform statistical analysis, cluster analysis and biochemical pathway analysis.

Biopsies from skeletal muscle and adipose tissue from both diabetics and nondiabetics will be applied. Changes in genes and biochemical pathways between diabetics and nondiabetics and functional relationships between adipose tissue and skeletal muscle will be investigated.

Grouping of subtypes in type 2 diabetes will be performed and a classification system will be constructed. Building a classifier may provide better and more precise diagnosis of type 2 diabetes.

Major advances in health science of type 2 diabetes thus seems to be promising and paving the way for individual treatment based on a more precise diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Of diabetic subjects:

* Type 2 diabetes
* Age: 30-65 years
* BMI: 27-35

Of nondiabetic subjects:

* Age: 30-65 years
* BMI: 27-35

Exclusion Criteria:

Of diabetic subjects:

* Medication, which have any influence on glucose metabolism and gene expression in adipose tissue and skeletal muscle at the time of sampling of biopsies.
* Disease in liver, heart, vessels or endocrine organs

Of nondiabetic subjects:

* Type 2 diabetes
* Relatives with type 2 diabetes
* Hyperglycemia
* Medication, which have any influence on glucose metabolism and gene expression in adipose tissue and skeletal muscle at the time of sampling of biopsies.
* Disease in liver, heart, vessels or endocrine organs

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-10; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Vibe Skov, MSc, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Clinical Biochemistry and Genetics, KKA, Odense C, Funen, Denmark